CLINICAL TRIAL: NCT07102615
Title: Intracervical Vasopressin for Completion of Hysteroscopic Removal of Retained Products of Conception
Brief Title: Intracervical Vasopressin
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2269142
Record Dates: First submitted 2025-07-31; First posted 2025-08-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Retained Products of Conception
Keywords: retained products of conception; intracervical; hysteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): Vasopressin- 20 mL of a dilute solution (5 units of Vasopressin in 20cc injectable saline)
  Interventions: Drug: Intracervical injection of Vasopressin
- Placebo (Placebo Comparator): 20 mL of saline
  Interventions: Drug: Intracervical Injection of saline

INTERVENTIONS:
Drug: Intracervical injection of Vasopressin — Intracervical injection of Vasopressin
  Arms: Treatment
Drug: Intracervical Injection of saline — Intracervical Injection of saline
  Arms: Placebo

SUMMARY:
This randomized study looks at whether using a medicine injected into the cervix of the uterus (intracervical), called vasopressin, helps to achieve better removal of retained products of conception (RPOC). RPOC means that after a pregnancy has ended (through miscarriage, abortion, or delivery), some parts of the pregnancy tissue, usually from the placenta or fetus, have stayed in the uterus. A hysteroscopic removal of RPOC is one type of treatment. This is a surgical procedure where a doctor uses a small camera attached to a thin tube (called a hysteroscope) to look inside the uterus.

The main goal of the study is :

• To add to the existing research through this study to see if the injection of intracervical vasopressin leads to improved completion rates of hysteroscopic management of RPOC.

Participants will:

• would be randomized to receive either vasopressin intracervical injection or a placebo injection (non-active saline) during your procedure. Information from the procedure will be collected from the participant's medical record.

DETAILED DESCRIPTION:
This double-blinded randomized control trial is designed to evaluate if intraoperative injection of intracervical vasopressin into the cervix will allow for completion of hysteroscopic removal of retained products of conception. This will be measured by surgical completion comparing patients who received intracervical vasopressin and those receiving placebo. Surgical completion is defined by completing the procedure without having to convert to suction of tissue due to bleeding or poor visualization. Secondary outcome measures include intraoperative bleeding, operative time, fluid deficit, and deficit volume.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Aged 18-51
* Undergoing surgical management for retained products of conception, postpartum retained products of conception or 1st trimester missed or incomplete abortion

Exclusion Criteria:

* Hemodynamic instability
* Active hemorrhage- soaking pad/hour
* Allergy to vasopressin
* Concern for intrauterine arteriovenous malformation
* Inability to consent

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Completion of procedure hysteroscopically | from start of procedure to end of procedure
  There is complete removal of RPOC hysteroscopically by the end of the procedure.

SECONDARY OUTCOMES:
Intraoperative Bleeding | from start of procedure to end of procedure
  calculated by dividing the number of red blood cells per milliliter of outflow distention fluid by the number of red blood cells per milliliter of the woman's blood immediately before the procedure and multiplying this quotient by the total amount of outflow fluid collected
Operative time | time from insertion of hysteroscope to procedure completion
  time from insertion of hysteroscope to procedure completion
fluid deficit volume | from start of procedure to end of procedure
  The difference between the total volume of distension fluid infusion into the uterine cavity during the hysteroscopy and the volume of fluid recovered from the outflow.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Miller, MD, Study Director — Prisma Health
Locations (1):
- The OB/GYN Center, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No